CLINICAL TRIAL: NCT04330534
Title: A Phase 1 Dose-ranging Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of BCX9930 in Healthy Subjects and in Subjects With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: First-in-Human Study of BCX9930 in Healthy Volunteers and Patients With PNH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX9930-101
Record Dates: First submitted 2020-03-23; First posted 2020-04-01 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Paroxysmal Nocturnal Hemoglobinuria; first-in-human; Factor D; complement inhibitor; alternative pathway inhibitor; BioCryst; proof-of-concept
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Intervention Model Description: Each cohort in Part 3 is enrolled as a single group; Parts 1 and 2 follow a parallel study model.
Masking Description: Part 3 is not masked; Parts 1 and 2 are participant and investigator masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCX9930 (Experimental): Parts 1, 2 and 3
  Interventions: Drug: BCX9930
- Placebo (Placebo Comparator): Parts 1 and 2 only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCX9930 — BCX9930 capsules for oral administration
  Arms: BCX9930
Drug: Placebo — placebo to match BCX9930 capsules for oral administration
  Arms: Placebo

SUMMARY:
This is a 3-part Phase 1 dose-ranging study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single (Part 1) and multiple (Part 2) ascending doses of BCX9930 in healthy subjects and in subjects with paroxysmal nocturnal hemoglobinuria (PNH; Part 3). Pharmacokinetics is an analysis of how the body handles the study drug BCX9930 and pharmacodynamics is an analysis of the activity that the study drug BCX9930 may have in the body.

DETAILED DESCRIPTION:
Up to 6 sequential ascending dose cohorts are planned to be dosed in a sequential manner in Part 1 of the study. Eight subjects will be treated with a single dose of the study drug per dose cohort (6 subjects per cohort will receive BCX9930 and 2 subjects per cohort will receive matching placebo). Escalation to the next higher dose level will occur only after completion of a review of clinical safety and pharmacokinetics by the Sponsor and PI.

Up to 7 ascending, multiple dose cohorts will be enrolled in a sequential manner in Part 2 of the study. In Cohorts 1 through 3, twelve subjects will be treated with either a 7-day or 14-day course of study drug (10 subjects per cohort will receive BCX9930 and 2 subjects per cohort will receive matching placebo) administered orally. In Cohorts 4 through 7, twelve subjects will be treated with a 3-day course of study drug (10 subjects per cohort will receive BCX9930 and 2 subjects per cohort will receive matching placebo) administered orally. The daily dose may be split into 2 times daily (BID) or 3 times daily (TID) dosing for the multiple ascending dose part as needed. Escalation to the next higher dose level in Part 2 will occur only after completion of a review of clinical safety and pharmacokinetics by the Sponsor and PI.

Part 3 of the study consists of up to 2 sequential ascending multiple dose cohorts of up to 8 subjects; each cohort may enroll up to 4 subjects with PNH who are naïve to both eculizumab and ravulizumab and up to 4 subjects with PNH who are currently being treated with either eculizumab or ravulizumab. In each cohort, subjects will receive one daily dose of BCX9930 on Days 1 to 14 and a higher daily dose on Days 15 to 28. Cohort 2 will start after independent data monitoring committee (DMC) review of Cohort 1 data and communication of their evaluation to Part 3 investigators. In South Africa, subjects that have clinical benefit from BCX9930 will be allowed to continue dosing for up to 48 weeks.

ELIGIBILITY:
Key Inclusion Criteria (Parts 1, 2, and 3):

* Able to provide written informed consent
* Acceptable birth control measures for male subjects and women of childbearing potential
* Is expected to adequately comply with required study procedures and restrictions

Key Inclusion Criteria (Parts 1 and 2):

* Body mass index (BMI) of 18.0 to 32.0 kg/m2.
* Males and non-pregnant, non-lactating females age 18 to 55 years.
* Part 2: Must have recent vaccination against Neisseria meningitidis and must be negative for colonisation by Neisseria meningitidis

Key Inclusion Criteria (Part 3 only):

* Male or non-pregnant, non-lactating female subjects ≥ 18 years old
* Have been diagnosed with PNH and have laboratory values indicative of active PNH
* Subjects naïve to both eculizumab and ravulizumab treatment, who have no access to, or are considered unsuitable for proven effective alternative options as per the local standard of care OR subjects currently receiving treatment with eculizumab or ravulizumab have been on a stable dose of eculizumab or ravulizumab for 6 months
* Must have recent vaccination against Neisseria meningitidis

Key Exclusion Criteria (Parts 1 and 2):

* Clinically significant medical history, current medical or psychiatric condition that, in the opinion of the Investigator or Sponsor, would interfere with the subject's ability to participate in the study or increase the risk of participation for that subject.
* Clinically significant ECG finding or laboratory/urinalysis abnormality
* Use of prescription or over the counter medication within 14 days of dosing
* Participation in any other investigational drug study within 90 days of screening
* Recent or current history of alcohol or drug abuse within the last 12 months
* Current smokers and those who have smoked within the last 12 months
* Positive serology for HIV or active infection with HBV or HCV
* Pregnant or nursing
* Donation or loss of greater than 400 mL of blood within 3 months
* History of severe hypersensitivity to any drug or Neisseria meningitidis vaccines (Part 2)
* Subject has recently received a live attenuated vaccine within 30 days of dosing or another type of vaccine within 14 days of Day 1

Key Exclusion Criteria (Part 3):

* Apart from a diagnosis of PNH, any clinically significant medical or psychiatric condition or medical history, other than those associated with PNH disease, that, in the opinion of the Investigator or Sponsor, would interfere with the subject's ability to participate in the study or participation would increase the risk for that subject
* Active bacterial infection
* Hereditary complement deficiency
* History of hematopoietic stem cell /marrow transplantation
* Current participation in any other investigational drug study or participation in an investigational drug study within 30 days of the screening visit
* History of meningococcal disease
* Positive drugs of abuse screen at screening visit
* Pregnant, planning to become pregnant, or having been pregnant within 90 days of Day 1, or lactating
* History of severe hypersensitivity to any drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 168 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Incidence of graded treatment-emergent adverse events | Part 1: Day 16
Incidence of graded treatment-emergent adverse events | Part 2: Day 23 (cohorts with 3 and 7 day dosing duration) or Day 31 (cohorts with 14 day dosing duration)
Incidence of graded treatment-emergent adverse events | Part 3:Day 44 or Week 50 (South Africa only)
Incidence of graded laboratory chemistry abnormalities | Part 1: Day 16
Incidence of graded laboratory chemistry abnormalities | Part 2: Day 23 (cohorts with 3 and 7 day dosing duration) or Day 31 (cohorts with 14 day dosing duration)
Incidence of graded laboratory chemistry abnormalities | Part 3:Day 44 or Week 50 (South Africa only)
Incidence of graded urinalysis abnormalities | Part 1: Day 16
Incidence of graded urinalysis abnormalities | Part 2: Day 23 (cohorts with 3 and 7 day dosing duration) or Day 31 (cohorts with 14 day dosing duration)
Incidence of graded urinalysis abnormalities | Part 3: Day 44 or Week 50 (South Africa only)
Incidence of graded coagulation abnormalities | Part 1: Day 16
Incidence of graded coagulation abnormalities | Part 2: Day 23 (cohorts with 3 and 7 day dosing duration) or Day 31 (cohorts with 14 day dosing duration)
Incidence of graded coagulation abnormalities | Part 3: Day 44 or Week 50 (South Africa only)
Incidence of graded hematology abnormalities | Part 1: Day 16
Incidence of graded hematology abnormalities | Part 2: Day 23 (cohorts with 3 and 7 day dosing duration) or Day 31 (cohorts with 14 day dosing duration)
Incidence of graded hematology abnormalities | Part 3: Day 44 or Week 50 (South Africa only)
Change from baseline in blood pressure | Part 1: Day 16
Change from baseline in blood pressure | Part 2: Day 23 (cohorts with 3 and 7 day dosing duration) or Day 31 (cohorts with 14 day dosing duration)
Change from baseline in blood pressure | Part 3: Day 44 or Week 50 (South Africa only)
Change from baseline in temperature | Part 1: Day 16
Change from baseline in temperature | Part 2: Day 23 (cohorts with 3 and 7 day dosing duration) or Day 31 (cohorts with 14 day dosing duration)
Change from baseline in temperature | Part 3: Day 44 or Week 50 (South Africa only)
Change from baseline in heart rate | Part 1: Day 16
Change from baseline in heart rate | Part 2: Day 23 (cohorts with 3 and 7 day dosing duration) or Day 31 (cohorts with 14 day dosing duration)
Change from baseline in heart rate | Part 3: Day 44 or Week 50 (South Africa only)
Change from baseline in respiratory rate | Part 3: Day 44 or Week 50 (South Africa only)
Change in Electrocardiogram (PR interval) | Part 1: Day 16
Change in Electrocardiogram (PR interval) | Part 2: Day 23 (cohorts with 3 and 7 day dosing duration) or Day 31 (cohorts with 14 day dosing duration)
Change in Electrocardiogram (PR interval) | Part 3: Day 44 or Week 50 (South Africa only)
Change in Electrocardiogram (QRS interval) | Part 1: Day 16
Change in Electrocardiogram (QRS interval) | Part 2: Day 23 (cohorts with 3 and 7 day dosing duration) or Day 31 (cohorts with 14 day dosing duration)
Change in Electrocardiogram (QRS interval) | Part 3: Day 44 or Week 50 (South Africa only)
Change in Electrocardiogram (RR interval) | Part 1: Day 16
Change in Electrocardiogram (RR interval) | Part 2: Day 23 (cohorts with 3 and 7 day dosing duration) or Day 31 (cohorts with 14 day dosing duration)
Change in Electrocardiogram (RR interval) | Part 3:Day 44 or Week 50 (South Africa only)
Change in Electrocardiogram (QT interval) | Part 1: Day 16
Change in Electrocardiogram (QT interval) | Part 2: Day 23 (cohorts with 3 and 7 day dosing duration) or Day 31 (cohorts with 14 day dosing duration)
Change in Electrocardiogram (QT interval) | Part 3:Day 44 or Week 50 (South Africa only)

SECONDARY OUTCOMES:
Plasma BCX9930 Cmax | plasma PK parameters are based on blood sampling through Day 4 for Part 1; through Day 6, 14 or 18 for Part 2 (Day depends on dosing duration); and through Day 28 for Part 3
Plasma BCX9930 Tmax | plasma PK parameters are based on blood sampling through Day 4 for Part 1; through Day 6, 14 or 18 for Part 2 (Day depends on dosing duration); and through Day 28 for Part 3
Plasma BCX9930 AUCinf | plasma PK parameters are based on blood sampling through Day 4 for Part 1
Plasma BCX9930 t1/2 | plasma PK parameters are based on blood sampling through Day 4 for Part 1; through Day 6, 14 or 18 for Part 2 (Day depends on dosing duration); and through Day 28 for Part 3
Plasma BCX9930 AUCtau | plasma PK parameters are based on blood sampling through Day 6, 14 or 18 for Part 2 (Day depends on dosing duration); and through Day 28 for Part 3
Serum AP complement activity | Part 1:through Study Day 4; through Day 6, 14 or 18 for Part 2 (Day depends on dosing duration); and Part 3 through Day 28 or Week 48 (South Africa only)
Plasma Factor Bb | Part 1:through Study Day 4; through Day 6, 14 or 18 for Part 2 (Day depends on dosing duration); and Part 3 through Day 28 or Week 48 (South Africa only)
Number of blood transfusions | Part 3:baseline through Day 28 or Week 50 (South Africa only)
Lactate dehydrogenase | Part 3: absolute and change from baseline through Day 28 or Week 50 (South Africa only)
Hemoglobin | Part 3: absolute and change from baseline through Day 28 or Week 50 (South Africa only)
Absolute reticulocyte count | Part 3: values and change from baseline through Day 28 or Week 50 (South Africa only)
Haptoglobin | Part 3: absolute and change from baseline through Day 28 or Week 50 (South Africa only)

CONTACTS AND LOCATIONS:
Overall Officials: Antionio Risitano, Principal Investigator — University of Naples
Locations (4):
- Study Site, Vienna, Austria
- South Africa (2):
  - Study Site, Bloemfontein
  - Study Site, Pretoria
- Study Site, London, United Kingdom